CLINICAL TRIAL: NCT04547699
Title: Impact of Cytokine Supplementation With Various Protein Concentrations Into Human in Vitro Culture Medium on ICSI Cycle Outcome
Brief Title: Cytokines Supplementation to Culture Media and ICSI Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Collaborators: Rahem Fertility Center (Other)
Responsible Party: Principal Investigator, Emad Mohamad Sedeek, Senior embryologist in IVF laboratory,, Mansoura Integrated Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cytokine plus Global Protein
Record Dates: First submitted 2020-08-30; First posted 2020-09-14 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: ICSI

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blinded and prospective study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSA (Placebo Comparator): A single step culture medium (SSCM; Global, Life Global)+5mg/ml (10% Vol/Vol) life global protein,
  Interventions: Combination Product: A single step culture medium
- CYK+ high HSA (Experimental): A single step culture medium (SSCM; Global, Life Global)+5mg/ml (10% Vol/Vol) life global protein, supplemented with 2ng/mL GM-CSF (G5035 Sigma), 5ng/mL HB-EGF (E4643 Sigma),and 5ng/mL LIF (SRP9001 Sigma).
  Interventions: Combination Product: A single step culture medium
- CYK+low HSA (Active Comparator): A single step culture medium (SSCM; Global, Life Global) +2mg/ml (5% Vol/Vol) life global protein, supplemented with 2ng/mL GM-CSF (G5035 Sigma), 5ng/mL HB-EGF (E4643 Sigma), and 5ng/mL LIF (SRP9001 Sigma).
  Interventions: Combination Product: A single step culture medium

INTERVENTIONS:
Combination Product: A single step culture medium — A single step culture medium (SSCM; Global, Life Global)+5mg/ml life global protein, without supplementation of CYK

SUMMARY:
A randomized clinical trial to evaluate the effect of cytokine supplementation in embryo culture medium with various protein concentrations aiming to evaluate the effects of cytokines (CYK) integration into the human in vitro culture medium with high and low human serum albumin (HSA) concentrations on live birth rates after intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
Oocytes were injected, and embryos cultured and transferred in three supplemented culture media.

A- A single step culture medium (SSCM; Global, Life Global)+5mg/ml (10% Vol/Vol), life global protein, without supplementation of CYK (control n=200), B- A single step culture medium (SSCM; Global, Life Global)+5mg/ml (10% Vol/Vol), life global protein, with 2ng/mL GM-CSF (granulocyte macrophage colony stimulating factor) (G5035 Sigma), 5ng/mL HB-EGF (Heparine Binding Epidermal Growth Factor )(E4643 Sigma),and 5ng/mL LIF (Lukemia Inhbitory Factor) (SRP9001 Sigma)(n=200).

C- A single step culture medium (SSCM; Global, Life Global) +2mg/ml (5% Vol/Vol) life global protein, with 2ng/mL GM-CSF (G5035 Sigma), 5ng/mL HB-EGF (E4643 Sigma), and 5ng/mL LIF (SRP9001 Sigma).(n=200) Setting :- - Mansoura Integrated Fertility

ELIGIBILITY:
Inclusion Criteria:

* Patients who fitted the medical definition of infertility "One year of unprotected intercourse but not pregnant".

Exclusion Criteria:

* History of ovarian or adnexal surgery.
* Suspicious findings of ovarian malignancy.
* Presence of endocrine disorders such as diabetes mellitus, hyper-prolactinemia, thyroid dysfunction, congenital adrenal hyperplasia, Cushing's syndrome, and adrenal insufficiency.
* Presence of Globozoospermia (100% round-headed spermatozoa)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 700 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
live birth rate | 9 months
  the number of deliveries that resulted in at least one live born baby (>20 weeks gestational age or 500 gm birth weight ) expressed per 100 embryo transfer,

SECONDARY OUTCOMES:
Fertilization rate | 4 weeks
  Fertilization rate (fertilized oocytes with two pronuclei/ number of MII oocytes) ×100 %
Top quality day 3 embryos | 4 weeks
  embryos with seven or eight blastomeres of stage-proper sizes, and <10% fragmentation by volume
Blastocyst formation rate | 4 weeks
  (number of blastocysts/number of cultured embryos for blastocyst formation) ×100%
Top blastocyst rate | 4 weeks
  (number of high quality blastocysts/number of formed blastocysts) ×100%
Available embryo rate | 4 weeks
  number of transferred and frozen embryos/number of zygotes (2 pronuclei) ×100%
clinical pregnancy rate | 8 weeks
  number of cycles with clinical pregnancy/number of transferred cycles) ×100%
Biochemical pregnancy rate | 6 weeks
  number of cycles with biochemical pregnancy/number of Cycles with positive HCG) ×100%.
Implantation rate | 8 weeks
  number of implanted embryos/number of transferred embryos) ×100%
Early embryo loss rat | 16 weeks
  number of early spontaneously aborted embryos/number of transferred embryos) × 100%.
ongoing pregnancy rate | 16 weeks
  number of clinical pregnancies after 12 weeks divided by number of embryo transfers multiplied by 100

CONTACTS AND LOCATIONS:
Overall Officials: Emad M Sedeek, MS, Principal Investigator — MIFC
Locations (2):
- Egypt (2):
  - Mansoura Integrated fertility Center, Al Mansurah, Dekahlia
  - Mansoura Integrated Fertility Center, Al Mansurah

IPD SHARING:
Plan to Share IPD: Yes
all IPD will be shared
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after completion and for 3 months

REFERENCES:
- [Background] Fukui Y, Hirota Y, Matsuo M, Gebril M, Akaeda S, Hiraoka T, Osuga Y. Uterine receptivity, embryo attachment, and embryo invasion: Multistep processes in embryo implantation. Reprod Med Biol. 2019 May 24;18(3):234-240. doi: 10.1002/rmb2.12280. eCollection 2019 Jul. PMID 31312101
- [Background] Guzeloglu-Kayisli O, Kayisli UA, Taylor HS. The role of growth factors and cytokines during implantation: endocrine and paracrine interactions. Semin Reprod Med. 2009 Jan;27(1):62-79. doi: 10.1055/s-0028-1108011. Epub 2009 Feb 5. PMID 19197806
- [Background] Fawzy M, Emad M, Elsuity MA, Mahran A, Abdelrahman MY, Fetih AN, Abdelghafar H, Sabry M, Nour M, Rasheed SM. Cytokines hold promise for human embryo culture in vitro: results of a randomized clinical trial. Fertil Steril. 2019 Nov;112(5):849-857.e1. doi: 10.1016/j.fertnstert.2019.07.012. Epub 2019 Sep 21. PMID 31551154